CLINICAL TRIAL: NCT04793594
Title: Tele-Assessment in Patients With Stroke: Which of the Berg Balance Scale, Tinetti Balance and Walk Test, Timed Up and Go Tests is More Effective in Balance Assessment?
Brief Title: Which Balance Test is More Effective When Evaluating Stroke Patients With a Tele-assessment?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ceren Bayrak, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC7
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Tele-assessment; Balance; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tele- Assessment Group: Balance Assessment
  Interventions: Other: Berg Balance Test; Other: Tinetti Balance And Gait Test; Other: Time Up And Go Test
- Face To Face (Clinic) Group: Balance Assessment
  Interventions: Other: Berg Balance Test; Other: Tinetti Balance And Gait Test; Other: Time Up And Go Test

INTERVENTIONS:
Other: Berg Balance Test — Patients evaluate with Berg Balance Test for balance
Other: Tinetti Balance And Gait Test — Patients evaluate with Tinetti Balance And Gait Test for balance
Other: Time Up And Go Test — Patients evaluate with Time Up And Go Test for balance

SUMMARY:
The aim of this study is to compare the feasibility levels and advantages of balance tests applied with tele-assessment methods to clinical application methods in stroke patients and to reveal their effectiveness.

DETAILED DESCRIPTION:
The aim of this study is to compare the feasibility levels and advantages of balance tests applied with tele-assessment methods to clinical application methods in stroke patients and to reveal their effectiveness. Stroke patients who are referred to İstinye University Bahçeşehir Liv Hospital Physiotherapy and Rehabilitation Unit at March-September for physiotherapy and meet the inclusion criteria will be included in the study. The Patient Assessment Form which were prepared by the researcher and the Standardized Mini Mental Test, The Rankin Scale, Timed Get Up and Go Test, Berg Balance Scale, Tinetti Balance and Gait Test in order to evaluate the balance and walking of the participants due to stroke and to compare the applicability level of the tests applied with the tele- assessment method and tests will be completed by individuals who agreed to participate in the study and / or the researchers who carried out the study.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient cognitive function for communication (Standardized Mini-Mental Test score> 24)
* Not dependent on bed or wheelchair. (1 ≤ Modified Rankin Scale score <5)
* Balance problem (Timed Get Up and Go Test score> 12 sec)
* Providing the necessary technological competence for remote video communication at home
* Near a relative who can accompany you during the assessment
* Age 20-80 years
* Speaking Turkish

Exclusion Criteria:

* Individuals with a neurological and orthopedic disease other than stroke, whose vision and auditory function are affected by stroke, and those with aphasia will not be included in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke is a serious life-threatening medical condition that happens when the blood supply to part of the brain is cut off.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Test | 12 weeks
  Berg Balance Test is consisting of 14 items and measures the ability of individuals to maintain balance while performing functional tasks. Each task is scored from 0 (cannot perform independently) to 4 (stated best performance). 0-20 points are interpreted as high risk of falling, between 21-40 points as medium risk of falling, and between 41-56 points as low risk. The validity and reliability study of the Turkish version in stroke patients was performed by Şahin et al.
Tinetti Balance And Gait Scale | 12 weeks
  Tinetti Balance And Gait Scale is a total of 28 points, with a maximum of 16 and a walking score of 12 points. Those who score 26 and below are thought to have problems; It is observed that the risk of self-falling is five times higher in those who score 19 and below compared to normal individuals (17). Its adaptation to Turkish, validity and reliability study was carried out by Ağırcan in 2009.
Timed Up And Go Test | 12 weeks
  Timed Up And Go Test is a simply and widely used and rapid test for assessing mobility and dinamic balance. The person is asked to stand up from the chair, walk 3 meters safely and at a normal pace, turn around, walk back, sit back on the chair, and the time is recorded in seconds (sec). The test is started with the patient's feet flat on the floor and arms resting on the armrest of the chair, and is performed in three repetitions and the best result is recorded. Walking longer than 12 seconds indicates a risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Bayrak, BSc, Principal Investigator — Istanbul University- Cerrahpasa, Faculty of Health Science, Physiotherapy And Rehabilitation Department; Ayse Zengin Alpozgen, PhD, Study Chair — Istanbul University- Cerrahpasa, Faculty of Health Science, Physiotherapy And Rehabilitation Department; Yakup Krespi, Professor, Principal Investigator — Istinye University, Faculty of Medicine, Neurology Department; Roya Soltanalizadeh, MD, Principal Investigator — Istinye University Bahcesehir Liv Hospital; İlknur Mazı, BSc, Principal Investigator — Istanbul University- Cerrahpasa, Faculty of Health Science, Physiotherapy And Rehabilitation Department